CLINICAL TRIAL: NCT03387150
Title: A Multicenter, Randomized, Partially Blinded Phase 1 Clinical Trial to Evaluate the Safety and Serum Concentrations of a Human Monoclonal Antibody, VRC-HIVMAB075-00-AB (VRC07-523LS), Administered in Multiple Doses and Routes to Healthy, HIV-uninfected Adults
Brief Title: Evaluating the Safety and Serum Concentrations of a Human Monoclonal Antibody, VRC-HIVMAB075-00-AB (VRC07-523LS), Administered in Multiple Doses and Routes to Healthy, HIV-uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 127/HPTN 087; 38458 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Results first posted 2022-03-21 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Group 1: VRC07-523LS (Experimental): Participants in Group 1 will receive 2.5 mg/kg of VRC07-523LS by IV infusion at Weeks 0, 16, 32, 48, and 64.
  Interventions: Biological: VRC07-523LS
- Group 2: VRC07-523LS (Experimental): Participants in Group 2 will receive 5 mg/kg of VRC07-523LS by IV infusion at Weeks 0, 16, 32, 48, and 64.
  Interventions: Biological: VRC07-523LS
- Group 3: VRC07-523LS (Experimental): Participants in Group 3 will receive 20 mg/kg of VRC07-523LS by IV infusion at Weeks 0, 16, 32, 48, and 64.
  Interventions: Biological: VRC07-523LS
- Group 4: VRC07-523LS (Experimental): Participants in Group 4 will receive 2.5 mg/kg of VRC07-523LS by SC injection at Weeks 0, 16, 32, 48, and 64.
  Interventions: Biological: VRC07-523LS
- Group 5: VRC07-523LS (Experimental): Participants in Group 5 will receive 5 mg/kg of VRC07-523LS by SC injection at Weeks 0, 16, 32, 48, and 64.
  Interventions: Biological: VRC07-523LS
- Group T6 VRC07-523LS (Experimental): Participants in Group T6 will receive 2.5 mg/kg of VRC07-523LS by IM injection at Weeks 0, 16, 32, 48, and 64.
  Interventions: Biological: VRC07-523LS
- Group P6: Placebo (Placebo Comparator): Participants in Group P6 will receive 2.5 mg/kg of placebo by IM injection at Weeks 0, 16, 32, 48, and 64.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: VRC07-523LS — Administered by intravenous (IV) infusion, subcutaneous (SC) injection, or intramuscular (IM) injection, depending on which group participants are in
  Other Names: VRC-HIVMAB075-00-AB
  Arms: Group 1: VRC07-523LS; Group 2: VRC07-523LS; Group 3: VRC07-523LS; Group 4: VRC07-523LS; Group 5: VRC07-523LS; Group T6 VRC07-523LS
Biological: Placebo — Sodium Chloride for Injection USP, 0.9%; administered by IM injection
  Arms: Group P6: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and serum concentrations of a human monoclonal antibody, VRC-HIVMAB075-00-AB (VRC07-523LS), administered in multiple doses and routes to healthy, HIV-uninfected adults.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability, and serum concentrations of a human monoclonal antibody, VRC-HIVMAB075-00-AB (VRC07-523LS), administered in multiple doses and routes to healthy, HIV-uninfected adults.

Participants will be randomly assigned to one of six groups. Participants in Group 1 will receive 2.5 mg/kg of VRC07-523LS by intravenous (IV) infusion at Weeks 0, 16, 32, 48, and 64. Participants in Group 2 will receive 5 mg/kg of VRC07-523LS by IV infusion at Weeks 0, 16, 32, 48, and 64. Participants in Group 3 will receive 20 mg/kg of VRC07-523LS by IV infusion at Weeks 0, 16, 32, 48, and 64. Participants in Group 4 will receive 2.5 mg/kg of VRC07-523LS by subcutaneous (SC) injection at Weeks 0, 16, 32, 48, and 64. Participants in Group 5 will receive 5 mg/kg of VRC07-523LS by SC injection at Weeks 0, 16, 32, 48, and 64. Participants in Group 6 will receive 2.5 mg/kg of VRC07-523LS or placebo by intramuscular (IM) injection at Weeks 0, 16, 32, 48, and 64.

Participants will attend numerous study visits throughout the course of the study, beginning at Week 0 through Week 112. Visits may include physical examinations, blood and urine collection, HIV testing, risk reduction counseling, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria

* Age of 18 to 50 years
* Access to a participating clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: volunteer demonstrates understanding of this study and completes a questionnaire prior to first study product administration with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Agrees not to enroll in another study of an investigational research agent until completion of the last required protocol clinic visit
* Good general health as shown by medical history, physical exam, and screening laboratory tests

HIV-Related Criteria:

* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling.
* Assessed by the clinic staff as being at 'low risk' for HIV infection and committed to maintaining behavior consistent with those criteria through the last required protocol clinic visit (see the protocol for more information).

Laboratory Inclusion Values

Hemogram/Complete Blood Count (CBC)

* Hemoglobin greater than or equal to 11.0 g/dL for volunteers who were assigned female sex at birth, greater than or equal to 13.0 g/dL for volunteers who were assigned male sex at birth. For transgender participants who have been on hormone therapy for more than 6 consecutive months, determine hemoglobin eligibility based on the gender with which they identify (ie, a transgender female who has been on hormone therapy for more than 6 consecutive months should be assessed for eligibility using the hemoglobin parameters for volunteers assigned female sex at birth).
* White blood cell (WBC) count equal to 2,500 to 12,000 cells/mm^3
* WBC differential either within institutional normal range or with site physician approval
* Platelets equal to 125,000 to 550,000/mm^3

Chemistry

* Chemistry panel: Alanine aminotransferase (ALT) less than 1.25 times the institutional upper limit of normal and creatinine less than or equal to institutional upper limits of normal.

Virology

* Negative HIV-1 and -2 blood test: US volunteers must have a negative US Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA) or chemiluminescent microparticle immunoassay (CMIA). Non-US sites may use locally available assays that have been approved by HVTN and HIV Prevention Trials Network (HPTN) Laboratory Operations.
* Negative Hepatitis B surface antigen (HBsAg)
* Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive

Urine

* Negative or trace urine protein

Reproductive Status

* Volunteers who were assigned female sex at birth: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to study product administration on the day of initial study infusion/injection. Persons who are NOT of reproductive potential due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.
* Reproductive status: A volunteer who was assigned female sex at birth must:

  * Agree to use effective contraception (see protocol for more information) for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit. Effective contraception is defined as using the following methods:
  * Condoms (male or female) with or without a spermicide,
  * Diaphragm or cervical cap with spermicide,
  * Intrauterine device (IUD),
  * Hormonal contraception, or
  * Any other contraceptive method approved by the HVTN 127/HPTN 087 Protocol Safety Review Team (PSRT)
  * Successful vasectomy in any partner assigned male sex at birth (considered successful if a volunteer reports that a partner assigned male sex at birth has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy);
  * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
  * Or plan to be sexually abstinent until at least 6 months following the last study product administration.
* Volunteers who were assigned female sex at birth must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion Criteria:

General

* Weight greater than 115 kg
* Blood products received within 120 days before first study product administration, unless eligibility for earlier enrollment is determined by the HVTN 127/HPTN 087 PSRT
* Investigational research agents received within 30 days before first study product administration
* Intent to participate in another study of an investigational research agent or any other study that requires non-Network HIV antibody testing during the planned duration of the HVTN 127/HPTN 087 study
* Pregnant or breastfeeding

Vaccines and other Injections

* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 127/HPTN 087 PSRT will determine eligibility on a case-by-case basis.
* Previous receipt of humanized or human mAbs, whether licensed or investigational; the HVTN 127/HPTN 087 PSRT will determine eligibility on a case-by-case basis.
* Previous receipt of monoclonal antibodies VRC01, VRC01LS, or VRC07-523LS

Immune System

* Immunosuppressive medications received within 30 days before first injection or infusion (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral prednisone or equivalent at doses less than 2 mg/kg/day and length of therapy less than 11 days with completion at least 30 days prior to enrollment)
* Serious adverse reactions to VRC07-523LS formulation components, including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain
* Immunoglobulin received within 90 days before first injection or infusion, unless eligibility for earlier enrollment is determined by the HVTN 127/HPTN 087 PSRT
* Autoimmune disease (Not excluded from participation: Volunteer with mild, stable and uncomplicated autoimmune disease that does not require immunosuppressive medication and that, in the judgment of the site investigator, is likely not subject to exacerbation and likely not to complicate Solicited and Unsolicited adverse event (AE) assessments)
* Immunodeficiency

Clinically significant medical conditions

* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response,
  * A process that would require medication that affects the immune response,
  * Any contraindication to repeated injections, infusions, or blood draws, including inability to establish venous access,
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
  * A condition or process (eg, chronic urticaria or recent injection or infusion with evidence of residual inflammation) for which signs or symptoms could be confused with reactions to the study product, or
  * Any condition specifically listed among the exclusion criteria.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or Solicited AEs, or a volunteer's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) therapy
* Asthma other than mild or moderate, well-controlled asthma. (Symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program (NAEPP) Expert Panel report). Exclude a volunteer who:

  * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
  * Uses high dose inhaled corticosteroids, or
  * In the past year has had either of the following:
  * Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids;
  * Needed emergency care, urgent care, hospitalization, or intubation for asthma.
* Diabetes mellitus type 1 or type 2 (Not excluded: type 2 cases controlled with diet alone or a history of isolated gestational diabetes.)
* Hypertension:

  * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be less than or equal to 150 mm Hg systolic and less than or equal to 100 mm Hg diastolic. For these volunteers, blood pressure must be less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic at enrollment.
  * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at enrollment or diastolic blood pressure greater than or equal to 100 mm Hg at enrollment.
* Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: History of seizure(s) within past three years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Walsh, Study Chair — Brigham and Women's Hospital; Cynthia Gay, Study Chair — University of North Carolina, Chapel Hill
Locations (7):
- United States (6):
  - Alabama CRS, Birmingham, Alabama
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Fenway Health (FH) CRS, Boston, Massachusetts
  - Columbia P&S CRS, New York, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
- Lausanne Vaccine and Immunotherapy Center CRS, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Walsh SR, Gay CL, Karuna ST, Hyrien O, Skalland T, Mayer KH, Sobieszczyk ME, Baden LR, Goepfert PA, Del Rio C, Pantaleo G, Andrew P, Karg C, He Z, Lu H, Paez CA, Baumblatt JAG, Polakowski LL, Chege W, Anderson MA, Janto S, Han X, Huang Y, Dumond J, Ackerman ME, McDermott AB, Flach B, Piwowar-Manning E, Seaton K, Tomaras GD, Montefiori DC, Gama L, Mascola JR; HVTN 127/HPTN 087 Study Team. Safety and pharmacokinetics of VRC07-523LS administered via different routes and doses (HVTN 127/HPTN 087): A Phase I randomized clinical trial. PLoS Med. 2024 Jun 24;21(6):e1004329. doi: 10.1371/journal.pmed.1004329. eCollection 2024 Jun. PMID 38913710

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Vaccine: VRC07-523LS IV-2.5 mg/kg wks(0,16,32,48,64)
- Group 2: Vaccine: VRC07-523LS IV-5 mg/kg wks(0,16,32,48,64)
- Group 3: Vaccine: VRC07-523LS IV-20 mg/kg wks(0,16,32,48,64)
- Group 4: Vaccine: VRC07-523LS SC-2.5 mg/kg wks(0,16,32,48,64)
- Group 5: Vaccine: VRC07-523LS SC-5 mg/kg wks(0,16,32,48,64)
- Group 6: Vaccine: VRC07-523LS IM-2.5 mg/kg wks(0,16,32,48,64)
- Group 7: Placebo: IM-0.9% Sodium Chloride wks(0,16,32,48,64)
Period: Overall Study
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine | Group 7: Placebo
Started | 19 | 19 | 21 | 21 | 20 | 21 | 3
Safety Population | 19 | 19 | 21 | 21 | 20 | 21 | 3
Completed | 13 | 16 | 16 | 14 | 14 | 14 | 3
Not Completed | 6 | 3 | 5 | 7 | 6 | 7 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 3 | 4 | 1 | 2 | 0
Not completed — Lost to Follow-up | 3 | 2 | 2 | 3 | 3 | 3 | 0
Not completed — Participant unable to adhere to visit | 0 | 1 | 0 | 0 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine | Group 7: Placebo | Total
Number analyzed (Participants) | 19 | 19 | 21 | 21 | 20 | 21 | 3 | 124
Age, Continuous [Median (Full Range); unit: years] | 30 [18 to 50] | 30 [18 to 48] | 23 [19 to 50] | 29 [20 to 49] | 27 [21 to 37] | 27 [19 to 43] | 31 [24 to 35] | 28 [18 to 50]
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18 - 20 years | 4 | 3 | 4 | 1 | 0 | 2 | 0 | 14
  21 - 30 years | 6 | 7 | 11 | 11 | 17 | 13 | 1 | 66
  31 - 40 years | 6 | 7 | 4 | 3 | 3 | 3 | 2 | 28
  41 - 50 years | 3 | 2 | 2 | 6 | 0 | 3 | 0 | 16
  Above 50 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 8 | 11 | 15 | 13 | 11 | 3 | 75
  Male | 5 | 11 | 10 | 6 | 7 | 10 | 0 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 5 | 2 | 0 | 2 | 0 | 12
  Not Hispanic or Latino | 19 | 16 | 16 | 19 | 20 | 19 | 3 | 112
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 3 | 0 | 1 | 1 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 4 | 2 | 5 | 6 | 6 | 0 | 28
  White | 12 | 10 | 13 | 10 | 11 | 12 | 3 | 71
  More than one race | 2 | 2 | 1 | 3 | 2 | 1 | 0 | 11
  Unknown or Not Reported | 0 | 2 | 2 | 3 | 0 | 1 | 0 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  USA | 19 | 19 | 21 | 21 | 20 | 21 | 3 | 124

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Pain and/or Tenderness
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017]. The maximum grade observed for each symptom over the time frame is presented
Time Frame: Measured through 3 days after each vaccine dose at Weeks 0, 16, 32, 48, 64
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine | Group 7: Placebo
Number analyzed (Participants) | 19 | 19 | 21 | 21 | 20 | 21 | 3
Participants
  None | 12 | 11 | 15 | 8 | 5 | 7 | 2
  Mild | 6 | 8 | 5 | 11 | 15 | 13 | 1
  Moderate | 1 | 0 | 1 | 2 | 0 | 1 | 0
  Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Erythema and/or Induration
Description: as for outcome 1
Time Frame: Measured through 3 days after each vaccine dose at Weeks 0, 16, 32, 48, 64
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine | Group 7: Placebo
Number analyzed (Participants) | 19 | 19 | 21 | 21 | 20 | 21 | 3
Participants
  Erythema/Redness: None | 14 | 15 | 16 | 7 | 7 | 19 | 3
  Erythema/Redness: Not gradable | 3 | 4 | 3 | 2 | 3 | 0 | 0
  Erythema/Redness: Gr 1: 2.5 - less than 5cm dim. | 0 | 0 | 1 | 2 | 2 | 0 | 0
  Erythema/Redness: Gr 1: 6.25 - less than 25cm^2 area | 1 | 0 | 0 | 4 | 3 | 2 | 0
  Erythema/Redness: Gr 2: 5 - less than 10cm dim. | 0 | 0 | 1 | 2 | 5 | 0 | 0
  Erythema/Redness: Gr 2: 25 - less than 100cm^2 area | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Erythema/Redness: Gr 3: >= 10cm dim. | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Erythema/Redness: Gr 3: >= 100cm^2 area | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Erythema/Redness: Gr 3: complications AE | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema/Redness: Gr 4: complications AE | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema/Redness: Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Induration/Swelling: None | 19 | 16 | 20 | 12 | 12 | 18 | 3
  Induration/Swelling: Not gradable | 0 | 3 | 1 | 2 | 6 | 2 | 0
  Induration/Swelling: Gr 1: 2.5 - less than 5cm dim. | 0 | 0 | 0 | 4 | 0 | 0 | 0
  Induration/Swelling: Gr 1: 6.25 - less than 25cm^2 area | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Induration/Swelling: Gr 2: 5 - less than 10cm dim. | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Induration/Swelling: Gr 2: 25 - less than 100cm^2 area | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Induration/Swelling: Gr 3: >= 10cm dim. | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Induration/Swelling: Gr 3: >= 100cm^2 area | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Induration/Swelling: Gr 3: complications AE | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Induration/Swelling: Gr 4: complications AE | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Induration/Swelling: Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema and/or Induration: None | 14 | 15 | 16 | 6 | 6 | 17 | 3
  Erythema and/or Induration: Not gradable | 3 | 4 | 3 | 2 | 4 | 2 | 0
  Erythema and/or Induration: Gr 1: 2.5 - less than 5cm dim. | 0 | 0 | 1 | 3 | 2 | 0 | 0
  Erythema and/or Induration: Gr 1: 6.25 - less than 25cm^2 area | 1 | 0 | 0 | 4 | 3 | 2 | 0
  Erythema and/or Induration: Gr 2: 5 - less than 10cm dim. | 0 | 0 | 1 | 2 | 4 | 0 | 0
  Erythema and/or Induration: Gr 2: 25 - less than 100cm^2 area | 1 | 0 | 0 | 1 | 1 | 0 | 0
  Erythema and/or Induration: Gr 3: >= 10cm dim. | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Erythema and/or Induration: Gr 3: >= 100cm^2 area | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Erythema and/or Induration: Gr 3: complications AE | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema and/or Induration: Gr 4: complications AE | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema and/or Induration: Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017]. The following symptoms are considered as systemic reactogenicity if the onset date was within the periods of assessment specified in the protocol: malaise and/or fatigue, myalgia, headache, nausea, vomiting, chills, arthralgia, and body temperature. The item Max. Systemic Symptoms is the maximum of the individual systemic reactogenicities excluding body temperature for a participant.
Time Frame: Measured through 3 days after each vaccine dose at Weeks 0, 16, 32, 48, 64
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine | Group 7: Placebo
Number analyzed (Participants) | 19 | 19 | 21 | 21 | 20 | 21 | 3
Participants
  Malaise and/or fatigue: None | 10 | 10 | 7 | 12 | 13 | 14 | 1
  Malaise and/or fatigue: Mild | 6 | 5 | 7 | 6 | 6 | 4 | 2
  Malaise and/or fatigue: Moderate | 3 | 4 | 5 | 3 | 1 | 3 | 0
  Malaise and/or fatigue: Severe | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 18 | 16 | 14 | 18 | 17 | 17 | 3
  Myalgia: Mild | 1 | 3 | 2 | 2 | 3 | 4 | 0
  Myalgia: Moderate | 0 | 0 | 4 | 1 | 0 | 0 | 0
  Myalgia: Severe | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Myalgia: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache: None | 13 | 11 | 4 | 12 | 16 | 13 | 2
  Headache: Mild | 4 | 6 | 12 | 6 | 4 | 7 | 1
  Headache: Moderate | 2 | 2 | 5 | 3 | 0 | 1 | 0
  Headache: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 15 | 15 | 17 | 16 | 18 | 18 | 2
  Nausea: Mild | 4 | 2 | 1 | 5 | 1 | 3 | 1
  Nausea: Moderate | 0 | 2 | 3 | 0 | 1 | 0 | 0
  Nausea: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: None | 19 | 17 | 13 | 20 | 18 | 20 | 2
  Chills: Mild | 0 | 1 | 5 | 1 | 2 | 1 | 1
  Chills: Moderate | 0 | 1 | 3 | 0 | 0 | 0 | 0
  Chills: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: None | 19 | 16 | 14 | 19 | 19 | 19 | 3
  Arthralgia: Mild | 0 | 3 | 4 | 1 | 1 | 2 | 0
  Arthralgia: Moderate | 0 | 0 | 2 | 1 | 0 | 0 | 0
  Arthralgia: Severe | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Arthralgia: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Facial flushing: None | 19 | 18 | 17 | 19 | 19 | 19 | 3
  Facial flushing: Mild | 0 | 1 | 4 | 2 | 1 | 2 | 0
  Facial flushing: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Facial flushing: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Facial flushing: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-exertional dyspnea: None | 19 | 18 | 19 | 21 | 19 | 21 | 3
  Non-exertional dyspnea: Mild | 0 | 1 | 2 | 0 | 1 | 0 | 0
  Non-exertional dyspnea: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-exertional dyspnea: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-exertional dyspnea: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-exertional tachycardia: None | 19 | 19 | 21 | 21 | 20 | 21 | 3
  Non-exertional tachycardia: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-exertional tachycardia: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-exertional tachycardia: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-exertional tachycardia: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unexplained diaphoresis: None | 19 | 19 | 19 | 20 | 19 | 21 | 3
  Unexplained diaphoresis: Mild | 0 | 0 | 2 | 1 | 1 | 0 | 0
  Unexplained diaphoresis: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unexplained diaphoresis: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unexplained diaphoresis: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Generalized Pruritus: None | 19 | 19 | 21 | 21 | 19 | 21 | 3
  Generalized Pruritus: Mild | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Generalized Pruritus: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Generalized Pruritus: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Generalized Pruritus: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urticaria: None | 19 | 19 | 21 | 21 | 20 | 21 | 3
  Urticaria: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urticaria: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urticaria: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urticaria: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: None | 8 | 5 | 4 | 10 | 11 | 8 | 1
  Max. Systemic Symptoms: Mild | 7 | 9 | 8 | 5 | 8 | 10 | 2
  Max. Systemic Symptoms: Moderate | 4 | 5 | 7 | 6 | 1 | 3 | 0
  Max. Systemic Symptoms: Severe | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: None | 17 | 18 | 18 | 21 | 20 | 20 | 3
  Temperature: Mild | 2 | 1 | 3 | 0 | 0 | 0 | 0
  Temperature: Moderate | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Temperature: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Chemistry and Hematology Laboratory Measures - Alanine Aminotransferase (ALT)
Description: For each local laboratory measure, summary statistics were presented by treatment group and timepoint for the overall population.
Time Frame: Measured during screening, Days 0, 56, 112, 168, 224, 280, 336, 392, 448, 504, 728
Population: 'Overall Number of Participants Analyzed' represents participants enrolled and eligible for laboratory assessment. Participants do not have laboratory assessments if they attended the visit but laboratory specimens were not collected, missed the scheduled visit, or terminated participation in the study prior to the scheduled visit.
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine | Group 7: Placebo
Number analyzed (Participants) | 19 | 19 | 21 | 21 | 20 | 21 | 3
U/L
  ALT (SGPT) (U/L)- Screening | 16 [11 to 21] | 16 [13 to 21] | 16 [12 to 21] | 14 [12 to 17] | 18 [10.5 to 20] | 13 [13 to 20] | 13 [12 to 16]
  ALT (SGPT) (U/L)- 0/Enrollment: number analyzed (Participants) | 19 | 19 | 21 | 20 | 20 | 21 | 3
  ALT (SGPT) (U/L)- 0/Enrollment | 14 [9 to 17] | 16 [12 to 17] | 19 [12 to 22] | 13.5 [10 to 21] | 13 [11.5 to 21.5] | 12 [10 to 20] | 17 [15 to 33]
  ALT (SGPT) (U/L)- 56: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 21 | 3
  ALT (SGPT) (U/L)- 56 | 15 [10 to 23] | 16 [12 to 21] | 15 [12.5 to 23] | 13 [10 to 21] | 15 [11 to 24] | 13 [11 to 23] | 31 [13 to 114]
  ALT (SGPT) (U/L)- 112: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 20 | 3
  ALT (SGPT) (U/L)- 112 | 16 [11 to 18] | 20 [13 to 23] | 13 [11.5 to 20.5] | 12 [12 to 18] | 16 [14 to 25] | 14 [10.5 to 20.5] | 19 [16 to 42]
  ALT (SGPT) (U/L)- 168: number analyzed (Participants) | 16 | 18 | 18 | 20 | 18 | 19 | 3
  ALT (SGPT) (U/L)- 168 | 13.5 [11 to 21] | 14.5 [13 to 23] | 15 [10 to 21] | 14 [10 to 24.5] | 16.5 [14 to 28] | 15 [12 to 23] | 19 [13 to 38]
  ALT (SGPT) (U/L)- 224: number analyzed (Participants) | 16 | 17 | 20 | 19 | 19 | 20 | 3
  ALT (SGPT) (U/L)- 224 | 18 [10.5 to 22.5] | 17 [13 to 21] | 15.5 [11.5 to 19.5] | 13 [11 to 25] | 14 [12 to 20] | 14.5 [12.5 to 19] | 17 [13 to 39]
  ALT (SGPT) (U/L)- 280: number analyzed (Participants) | 14 | 17 | 17 | 19 | 19 | 19 | 2
  ALT (SGPT) (U/L)- 280 | 16 [10 to 29] | 18 [14 to 25] | 15 [13 to 20] | 15 [11 to 23] | 17 [11 to 22] | 14 [11 to 23] | 18 [14 to 22]
  ALT (SGPT) (U/L)- 336: number analyzed (Participants) | 15 | 17 | 18 | 19 | 16 | 17 | 3
  ALT (SGPT) (U/L)- 336 | 15 [11 to 23] | 17 [15 to 18] | 14.5 [11 to 22] | 15 [11 to 20] | 16 [11.5 to 20] | 15 [13 to 18] | 13 [11 to 41]
  ALT (SGPT) (U/L)- 392: number analyzed (Participants) | 14 | 15 | 17 | 18 | 17 | 17 | 3
  ALT (SGPT) (U/L)- 392 | 17 [10 to 34] | 16 [12 to 21] | 19 [11 to 23] | 15 [10 to 24] | 16 [14 to 28] | 15 [12 to 17] | 18 [14 to 39]
  ALT (SGPT) (U/L)- 448: number analyzed (Participants) | 13 | 16 | 16 | 17 | 15 | 17 | 3
  ALT (SGPT) (U/L)- 448 | 13 [11 to 20] | 16.5 [13.5 to 20.5] | 17.5 [13 to 19.5] | 16 [10 to 22] | 18 [11 to 32] | 13 [11 to 18] | 16 [14 to 38]
  ALT (SGPT) (U/L)- 504: number analyzed (Participants) | 12 | 16 | 12 | 16 | 12 | 17 | 3
  ALT (SGPT) (U/L)- 504 | 12 [9 to 16] | 15 [12.5 to 31] | 13.5 [11 to 16.5] | 14.5 [10 to 22] | 16.5 [10 to 20.5] | 17 [12 to 21] | 15 [11 to 53]
  ALT (SGPT) (U/L)- 728: number analyzed (Participants) | 1 | 7 | 4 | 6 | 4 | 4 | 1
  ALT (SGPT) (U/L)- 728 | 19 [19 to 19] | 16 [15 to 26] | 16 [13 to 28.5] | 18.5 [15 to 20] | 18 [12.5 to 25] | 14 [9 to 26] | 26 [26 to 26]

5. Primary Outcome: Chemistry and Hematology Laboratory Measures - Creatinine
Description: as for outcome 4
Time Frame: Measured during screening, Days 0, 56, 112, 168, 224, 280, 336, 392, 448, 504, 728
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine | Group 7: Placebo
Number analyzed (Participants) | 19 | 19 | 21 | 21 | 20 | 21 | 3
mg/dL
  Creatinine (mg/dL)- Screening | 0.85 [0.69 to 1] | 0.92 [0.78 to 1] | 0.84 [0.76 to 0.96] | 0.79 [0.7 to 0.9] | 0.84 [0.77 to 0.91] | 0.86 [0.72 to 0.98] | 0.74 [0.66 to 0.78]
  Creatinine (mg/dL)- 0/Enrollment: number analyzed (Participants) | 19 | 19 | 21 | 20 | 19 | 21 | 3
  Creatinine (mg/dL)- 0/Enrollment | 0.8 [0.76 to 1.05] | 0.93 [0.81 to 1] | 0.83 [0.72 to 0.93] | 0.83 [0.78 to 1.02] | 0.8 [0.65 to 0.9] | 0.83 [0.71 to 0.93] | 0.77 [0.64 to 0.81]
  Creatinine (mg/dL)- 56: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 21 | 3
  Creatinine (mg/dL)- 56 | 0.84 [0.7 to 1] | 0.9 [0.8 to 0.98] | 0.94 [0.75 to 1.02] | 0.82 [0.74 to 0.91] | 0.82 [0.68 to 1] | 0.8 [0.74 to 0.97] | 0.7 [0.66 to 0.74]
  Creatinine (mg/dL)- 112: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 20 | 3
  Creatinine (mg/dL)- 112 | 0.8 [0.69 to 0.89] | 0.88 [0.79 to 0.94] | 0.88 [0.71 to 1.02] | 0.86 [0.76 to 0.93] | 0.79 [0.7 to 0.96] | 0.84 [0.74 to 0.96] | 0.72 [0.64 to 0.75]
  Creatinine (mg/dL)- 168: number analyzed (Participants) | 16 | 18 | 18 | 20 | 18 | 19 | 3
  Creatinine (mg/dL)- 168 | 0.86 [0.75 to 0.92] | 0.91 [0.8 to 1] | 0.81 [0.73 to 0.93] | 0.83 [0.77 to 1] | 0.81 [0.7 to 0.95] | 0.9 [0.75 to 1] | 0.7 [0.68 to 0.79]
  Creatinine (mg/dL)- 224: number analyzed (Participants) | 16 | 17 | 20 | 19 | 19 | 20 | 3
  Creatinine (mg/dL)- 224 | 0.79 [0.69 to 0.9] | 0.86 [0.72 to 0.99] | 0.81 [0.72 to 0.95] | 0.81 [0.77 to 0.89] | 0.83 [0.67 to 0.94] | 0.82 [0.73 to 0.97] | 0.72 [0.68 to 0.8]
  Creatinine (mg/dL)- 280: number analyzed (Participants) | 14 | 17 | 17 | 19 | 19 | 19 | 2
  Creatinine (mg/dL)- 280 | 0.81 [0.71 to 0.88] | 0.89 [0.77 to 1.07] | 0.78 [0.72 to 0.95] | 0.81 [0.76 to 0.95] | 0.85 [0.7 to 0.9] | 0.89 [0.73 to 0.96] | 0.72 [0.7 to 0.74]
  Creatinine (mg/dL)- 336: number analyzed (Participants) | 15 | 17 | 18 | 19 | 16 | 17 | 3
  Creatinine (mg/dL)- 336 | 0.84 [0.69 to 0.9] | 0.85 [0.76 to 0.99] | 0.85 [0.72 to 0.93] | 0.84 [0.77 to 0.95] | 0.87 [0.77 to 1.01] | 0.87 [0.77 to 0.99] | 0.78 [0.7 to 0.89]
  Creatinine (mg/dL)- 392: number analyzed (Participants) | 14 | 15 | 17 | 18 | 17 | 17 | 3
  Creatinine (mg/dL)- 392 | 0.88 [0.7 to 0.9] | 0.95 [0.8 to 1.02] | 0.82 [0.8 to 0.96] | 0.85 [0.72 to 0.96] | 0.89 [0.76 to 1] | 0.89 [0.8 to 1] | 0.75 [0.71 to 0.9]
  Creatinine (mg/dL)- 448: number analyzed (Participants) | 13 | 16 | 16 | 17 | 15 | 17 | 3
  Creatinine (mg/dL)- 448 | 0.82 [0.76 to 0.91] | 0.9 [0.81 to 1] | 0.8 [0.72 to 0.91] | 0.81 [0.74 to 0.96] | 0.9 [0.74 to 0.97] | 0.84 [0.75 to 0.97] | 0.75 [0.7 to 0.76]
  Creatinine (mg/dL)- 504: number analyzed (Participants) | 12 | 16 | 12 | 16 | 12 | 17 | 3
  Creatinine (mg/dL)- 504 | 0.87 [0.76 to 1.06] | 0.92 [0.78 to 1.08] | 0.78 [0.71 to 0.98] | 0.85 [0.78 to 0.95] | 0.8 [0.72 to 0.86] | 0.88 [0.7 to 0.99] | 0.81 [0.7 to 0.84]
  Creatinine (mg/dL)- 728: number analyzed (Participants) | 1 | 7 | 4 | 6 | 4 | 4 | 1
  Creatinine (mg/dL)- 728 | 1.1 [1.1 to 1.1] | 1.1 [0.96 to 1.15] | 0.77 [0.68 to 0.92] | 0.87 [0.8 to 1.14] | 0.81 [0.77 to 0.86] | 0.89 [0.78 to 0.92] | 0.66 [0.66 to 0.66]

6. Primary Outcome: Chemistry and Hematology Laboratory Measures - Hemoglobin
Description: as for outcome 4
Time Frame: Measured during screening, Days 0, 56, 112, 168, 224, 280, 336, 392, 448, 504, 728
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine | Group 7: Placebo
Number analyzed (Participants) | 19 | 19 | 21 | 21 | 20 | 21 | 3
g/dL
  Hemoglobin (g/dL)- Screening | 13.3 [12.7 to 14] | 14.2 [13.5 to 15.3] | 13.8 [13.3 to 14.8] | 13.1 [12.7 to 14.1] | 13.8 [13.15 to 15.1] | 14.4 [13 to 15.2] | 13.4 [12.1 to 14.1]
  Hemoglobin (g/dL)- 0/Enrollment: number analyzed (Participants) | 19 | 19 | 21 | 20 | 20 | 21 | 3
  Hemoglobin (g/dL)- 0/Enrollment | 13.1 [12.3 to 14.2] | 13.9 [12.6 to 14.7] | 13.8 [12.8 to 14.5] | 13 [12.25 to 13.7] | 13.55 [13 to 15.2] | 14.1 [12.6 to 15] | 12.5 [11.7 to 13.4]
  Hemoglobin (g/dL)- 56: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 21 | 3
  Hemoglobin (g/dL)- 56 | 13.35 [12.7 to 13.8] | 14.25 [13.6 to 15.1] | 13.4 [12.45 to 14.85] | 12.9 [12.5 to 13.9] | 13.8 [12.8 to 14.6] | 14.4 [12 to 14.9] | 12.6 [12 to 13.1]
  Hemoglobin (g/dL)- 112: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 20 | 3
  Hemoglobin (g/dL)- 112 | 12.7 [11.9 to 13.9] | 13.95 [13.1 to 14.7] | 13.6 [12.55 to 15.15] | 13.1 [12.4 to 13.7] | 13.7 [12.6 to 14.6] | 14.45 [13.1 to 15.2] | 12.6 [12.2 to 14.1]
  Hemoglobin (g/dL)- 168: number analyzed (Participants) | 16 | 18 | 18 | 20 | 18 | 19 | 3
  Hemoglobin (g/dL)- 168 | 13.7 [12.65 to 14.75] | 14.1 [13 to 14.8] | 13.65 [13.1 to 15.5] | 13.25 [12.05 to 13.85] | 13.5 [13 to 14.7] | 14.5 [12.4 to 15.1] | 12.8 [12.3 to 13.8]
  Hemoglobin (g/dL)- 224: number analyzed (Participants) | 16 | 17 | 20 | 19 | 19 | 20 | 3
  Hemoglobin (g/dL)- 224 | 12.95 [12.3 to 13.8] | 13.7 [12.9 to 14.8] | 13.2 [12.5 to 14.95] | 13.5 [11.9 to 14.2] | 13.6 [13.3 to 14.7] | 14.15 [12.3 to 15] | 13.1 [11.8 to 13.3]
  Hemoglobin (g/dL)- 280: number analyzed (Participants) | 14 | 17 | 17 | 19 | 18 | 19 | 2
  Hemoglobin (g/dL)- 280 | 13.3 [12.6 to 14] | 13.7 [13.1 to 14.4] | 13.1 [12.9 to 14.7] | 13.3 [12.1 to 14.3] | 13.6 [12.9 to 14.6] | 14.2 [11.8 to 14.9] | 13.3 [12.2 to 14.4]
  Hemoglobin (g/dL)- 336: number analyzed (Participants) | 15 | 17 | 18 | 19 | 16 | 17 | 3
  Hemoglobin (g/dL)- 336 | 13.3 [12.5 to 14.4] | 13.6 [12.4 to 14.8] | 13.3 [12.3 to 15] | 13.3 [12.5 to 14.2] | 13.5 [12.75 to 15.2] | 14.2 [13.4 to 15.1] | 12.9 [12.2 to 13.5]
  Hemoglobin (g/dL)- 392: number analyzed (Participants) | 14 | 15 | 17 | 18 | 17 | 17 | 3
  Hemoglobin (g/dL)- 392 | 13.3 [12.4 to 14.2] | 14.2 [13.2 to 14.8] | 13.5 [12.6 to 15.3] | 13.4 [12.5 to 14.3] | 13.5 [13 to 14.7] | 14.3 [12.6 to 14.9] | 12.6 [12.6 to 14.9]
  Hemoglobin (g/dL)- 448: number analyzed (Participants) | 13 | 16 | 16 | 17 | 15 | 17 | 3
  Hemoglobin (g/dL)- 448 | 12.9 [12.5 to 13.5] | 13.95 [12.85 to 14.55] | 13.3 [12.2 to 14.4] | 13.3 [12.3 to 13.9] | 13.6 [12.7 to 14.8] | 14.2 [12.3 to 14.9] | 13 [11.9 to 13.7]
  Hemoglobin (g/dL)- 504: number analyzed (Participants) | 12 | 16 | 12 | 16 | 12 | 17 | 3
  Hemoglobin (g/dL)- 504 | 13.25 [12.3 to 14.05] | 14.35 [13.2 to 14.8] | 13.4 [12.6 to 13.9] | 13 [12.4 to 14.6] | 13.9 [12.85 to 14.75] | 14.4 [13.2 to 15.6] | 12.9 [12.1 to 14]
  Hemoglobin (g/dL)- 728: number analyzed (Participants) | 1 | 7 | 4 | 6 | 4 | 4 | 1
  Hemoglobin (g/dL)- 728 | 12.7 [12.7 to 12.7] | 14.7 [13.4 to 15] | 13.1 [12.45 to 14.55] | 14.9 [12.8 to 15.4] | 14.6 [13.65 to 15.5] | 14 [12.65 to 15.05] | 12.5 [12.5 to 12.5]

7. Primary Outcome: Chemistry and Hematology Laboratory Measures - Lymphocyte Count, Neutrophil Count
Description: as for outcome 4
Time Frame: Measured during screening, Days 0, 56, 112, 168, 224, 280, 336, 392, 448, 504, 728
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: 1000 cells /cubic mm
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine | Group 7: Placebo
Number analyzed (Participants) | 19 | 19 | 21 | 21 | 20 | 21 | 3
1000 cells /cubic mm
  Neutrophils (1000/cubic mm)- Screening | 3.84 [2.6 to 5] | 3.7 [2.95 to 4.15] | 3.72 [2.8 to 4.19] | 3.24 [2.7 to 3.93] | 3.76 [2.77 to 5.19] | 2.82 [2.3 to 4.51] | 3.37 [3.3 to 7.32]
  Neutrophils (1000/cubic mm)- 0/Enrollment: number analyzed (Participants) | 19 | 19 | 21 | 20 | 20 | 21 | 3
  Neutrophils (1000/cubic mm)- 0/Enrollment | 2.95 [2.49 to 4.67] | 4.01 [3.16 to 4.73] | 3.92 [2.62 to 4.95] | 2.98 [2.3 to 3.97] | 3.31 [2.92 to 4.17] | 3.16 [2.42 to 3.94] | 5.82 [2.98 to 6.61]
  Neutrophils (1000/cubic mm)- 56: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 21 | 3
  Neutrophils (1000/cubic mm)- 56 | 3.12 [2.18 to 3.8] | 3.83 [3.02 to 4.94] | 4 [2.84 to 4.61] | 2.78 [2.4 to 4.06] | 3.47 [2.74 to 4.2] | 3.28 [2.27 to 4.07] | 7.27 [6.07 to 7.95]
  Neutrophils (1000/cubic mm)- 112: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 20 | 3
  Neutrophils (1000/cubic mm)- 112 | 3.65 [3 to 4.07] | 3.87 [3.25 to 4.61] | 3.89 [2.8 to 5.28] | 3.03 [2.4 to 3.35] | 3.02 [2.62 to 3.61] | 3.17 [2.5 to 4.1] | 5.9 [4.9 to 6.6]
  Neutrophils (1000/cubic mm)- 168: number analyzed (Participants) | 16 | 18 | 18 | 20 | 18 | 19 | 3
  Neutrophils (1000/cubic mm)- 168 | 3.35 [2.07 to 4.77] | 3.1 [2.66 to 3.87] | 3.61 [2.65 to 4.35] | 3.17 [2.68 to 4.42] | 3.19 [2.75 to 4.06] | 2.84 [2.4 to 4.2] | 6.19 [4.85 to 7.03]
  Neutrophils (1000/cubic mm)- 224: number analyzed (Participants) | 15 | 17 | 20 | 18 | 19 | 20 | 3
  Neutrophils (1000/cubic mm)- 224 | 2.94 [1.95 to 3.82] | 3.55 [2.66 to 3.9] | 3.53 [2.73 to 4.29] | 2.89 [2.33 to 3.66] | 3.02 [2.44 to 3.7] | 2.75 [2.31 to 3.53] | 4.96 [4.85 to 6.87]
  Neutrophils (1000/cubic mm)- 280: number analyzed (Participants) | 14 | 17 | 17 | 19 | 18 | 19 | 2
  Neutrophils (1000/cubic mm)- 280 | 2.69 [2.02 to 3.9] | 3.64 [2.7 to 4.72] | 3.57 [2.98 to 4.6] | 3.12 [2.5 to 4.06] | 3.15 [2.53 to 4.83] | 2.94 [2.21 to 3.72] | 5.27 [4.54 to 5.99]
  Neutrophils (1000/cubic mm)- 336: number analyzed (Participants) | 15 | 17 | 18 | 19 | 16 | 17 | 3
  Neutrophils (1000/cubic mm)- 336 | 3.06 [2.2 to 4.69] | 3.55 [2.5 to 3.99] | 4.17 [3.14 to 4.52] | 3.04 [2.3 to 3.59] | 3.08 [2.33 to 3.66] | 2.83 [2.46 to 3.47] | 6.51 [5 to 7.58]
  Neutrophils (1000/cubic mm)- 392: number analyzed (Participants) | 14 | 15 | 17 | 18 | 17 | 17 | 3
  Neutrophils (1000/cubic mm)- 392 | 3.13 [2.34 to 4.34] | 3.61 [2.86 to 4.26] | 3.69 [2.85 to 4.27] | 2.86 [2.51 to 3.5] | 3.53 [2.7 to 3.94] | 2.84 [2.42 to 3.75] | 6.13 [5.04 to 7.56]
  Neutrophils (1000/cubic mm)- 448: number analyzed (Participants) | 13 | 16 | 16 | 17 | 15 | 17 | 3
  Neutrophils (1000/cubic mm)- 448 | 3.11 [2.34 to 4.16] | 3.76 [2.75 to 4.9] | 3.74 [3.14 to 5.09] | 3.05 [2.5 to 3.89] | 2.97 [2.18 to 4.47] | 3.04 [2.24 to 4.24] | 6.24 [5.09 to 6.46]
  Neutrophils (1000/cubic mm)- 504: number analyzed (Participants) | 12 | 16 | 12 | 16 | 12 | 17 | 3
  Neutrophils (1000/cubic mm)- 504 | 3.38 [1.97 to 3.66] | 3.86 [2.8 to 4.59] | 3.91 [2.53 to 5.81] | 2.81 [2.39 to 3.44] | 3.39 [2.72 to 3.71] | 3.02 [2.1 to 3.65] | 6.42 [4.95 to 8.12]
  Neutrophils (1000/cubic mm)- 728: number analyzed (Participants) | 1 | 7 | 4 | 5 | 4 | 4 | 1
  Neutrophils (1000/cubic mm)- 728 | 4.56 [4.56 to 4.56] | 4.25 [2.7 to 4.95] | 4.02 [3.25 to 5.21] | 2.3 [2.2 to 2.6] | 2.93 [2.45 to 3.78] | 3.63 [3.13 to 4.64] | 4.8 [4.8 to 4.8]
  Lymphocytes (1000/cubic mm)- Screening | 2 [1.64 to 2.4] | 1.98 [1.7 to 2.44] | 2.04 [1.48 to 2.14] | 1.6 [1.4 to 2.07] | 1.92 [1.71 to 2.26] | 1.86 [1.66 to 2.67] | 3.06 [2.14 to 3.25]
  Lymphocytes (1000/cubic mm)- 0/Enrollment: number analyzed (Participants) | 19 | 19 | 21 | 20 | 20 | 21 | 3
  Lymphocytes (1000/cubic mm)- 0/Enrollment | 1.86 [1.72 to 2.1] | 1.85 [1.6 to 2.25] | 1.87 [1.56 to 2.04] | 1.64 [1.44 to 2.21] | 1.86 [1.63 to 2.23] | 1.95 [1.55 to 2.29] | 2.94 [2.22 to 3.22]
  Lymphocytes (1000/cubic mm)- 56: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 21 | 3
  Lymphocytes (1000/cubic mm)- 56 | 1.98 [1.57 to 2.25] | 1.94 [1.56 to 2.11] | 1.99 [1.33 to 2.5] | 1.86 [1.55 to 2] | 2.12 [1.78 to 2.48] | 1.87 [1.68 to 2.44] | 2.97 [2.05 to 3.38]
  Lymphocytes (1000/cubic mm)- 112: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 20 | 3
  Lymphocytes (1000/cubic mm)- 112 | 1.82 [1.59 to 2.07] | 1.8 [1.5 to 2.24] | 2.04 [1.55 to 2.46] | 1.77 [1.4 to 2.03] | 1.91 [1.76 to 2.16] | 1.93 [1.51 to 2.36] | 3.46 [2.34 to 3.55]
  Lymphocytes (1000/cubic mm)- 168: number analyzed (Participants) | 16 | 18 | 18 | 20 | 18 | 19 | 3
  Lymphocytes (1000/cubic mm)- 168 | 1.76 [1.53 to 1.99] | 1.8 [1.53 to 1.96] | 1.86 [1.53 to 2.07] | 1.61 [1.31 to 1.97] | 1.97 [1.65 to 2.26] | 1.89 [1.4 to 2.33] | 3.27 [2.17 to 3.33]
  Lymphocytes (1000/cubic mm)- 224: number analyzed (Participants) | 15 | 17 | 20 | 18 | 19 | 20 | 3
  Lymphocytes (1000/cubic mm)- 224 | 1.65 [1.44 to 2.12] | 1.91 [1.6 to 2.1] | 2.01 [1.68 to 2.51] | 1.61 [1.41 to 1.99] | 1.94 [1.68 to 2.23] | 1.74 [1.49 to 2.37] | 3.13 [1.91 to 3.85]
  Lymphocytes (1000/cubic mm)- 280: number analyzed (Participants) | 14 | 17 | 17 | 19 | 18 | 19 | 2
  Lymphocytes (1000/cubic mm)- 280 | 1.93 [1.75 to 2.13] | 1.71 [1.59 to 2.1] | 1.73 [1.3 to 2.32] | 1.7 [1.4 to 1.9] | 2.1 [1.81 to 2.66] | 1.92 [1.78 to 2.54] | 2.86 [2.15 to 3.58]
  Lymphocytes (1000/cubic mm)- 336: number analyzed (Participants) | 15 | 17 | 18 | 19 | 16 | 17 | 3
  Lymphocytes (1000/cubic mm)- 336 | 2 [1.62 to 2.06] | 1.69 [1.5 to 2.05] | 2.16 [1.63 to 3.01] | 1.76 [1.21 to 2.18] | 2.12 [1.81 to 2.41] | 1.82 [1.54 to 2.21] | 2.95 [1.79 to 3.82]
  Lymphocytes (1000/cubic mm)- 392: number analyzed (Participants) | 14 | 15 | 17 | 18 | 17 | 17 | 3
  Lymphocytes (1000/cubic mm)- 392 | 1.79 [1.53 to 2.08] | 1.8 [1.51 to 2.1] | 2.01 [1.43 to 2.85] | 1.58 [1.38 to 1.93] | 1.91 [1.7 to 2.3] | 1.82 [1.39 to 2.3] | 2.82 [1.46 to 3.1]
  Lymphocytes (1000/cubic mm)- 448: number analyzed (Participants) | 13 | 16 | 16 | 17 | 15 | 17 | 3
  Lymphocytes (1000/cubic mm)- 448 | 1.89 [1.68 to 2] | 1.83 [1.52 to 2.11] | 1.96 [1.34 to 2.44] | 1.8 [1.4 to 1.96] | 1.89 [1.63 to 2.39] | 1.99 [1.44 to 2.31] | 2.87 [1.94 to 3.52]
  Lymphocytes (1000/cubic mm)- 504: number analyzed (Participants) | 12 | 16 | 12 | 16 | 12 | 17 | 3
  Lymphocytes (1000/cubic mm)- 504 | 1.92 [1.54 to 2.28] | 1.89 [1.65 to 2.12] | 1.84 [1.5 to 2.26] | 1.79 [1.42 to 2.09] | 1.94 [1.85 to 2.29] | 1.76 [1.4 to 2.3] | 2.96 [1.3 to 3.02]
  Lymphocytes (1000/cubic mm)- 728: number analyzed (Participants) | 1 | 7 | 4 | 5 | 4 | 4 | 1
  Lymphocytes (1000/cubic mm)- 728 | 1.85 [1.85 to 1.85] | 1.7 [1.5 to 1.95] | 2.24 [1.79 to 3] | 1.5 [1.4 to 1.51] | 2.65 [1.95 to 3.45] | 1.69 [1.52 to 2.03] | 3.89 [3.89 to 3.89]

8. Primary Outcome: Chemistry and Hematology Laboratory Measures - Platelets, White Blood Cells (WBC)
Description: as for outcome 4
Time Frame: Measured during screening, Days 0, 56, 112, 168, 224, 280, 336, 392, 448, 504, 728
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: 1000 cells/cubic mm
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine | Group 7: Placebo
Number analyzed (Participants) | 19 | 19 | 21 | 21 | 20 | 21 | 3
1000 cells/cubic mm
  WBC (1000/cubic mm)- Screening | 6.4 [5 to 7.8] | 6.15 [5.36 to 7.44] | 6.8 [5.1 to 7.6] | 6.06 [4.54 to 6.59] | 6.7 [5.08 to 7.6] | 5.9 [4.71 to 8.5] | 7.1 [5.9 to 11.4]
  WBC (1000/cubic mm)- 0/Enrollment: number analyzed (Participants) | 19 | 19 | 21 | 20 | 20 | 21 | 3
  WBC (1000/cubic mm)- 0/Enrollment | 6.2 [4.7 to 7.37] | 6.9 [5.4 to 7.7] | 6.51 [4.9 to 7.5] | 5.65 [4.56 to 6.43] | 6.1 [5.56 to 6.85] | 5.9 [4.73 to 6.79] | 9.8 [5.7 to 10.2]
  WBC (1000/cubic mm)- 56: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 21 | 3
  WBC (1000/cubic mm)- 56 | 5.41 [4.6 to 7.1] | 6.76 [5.5 to 7.69] | 6.45 [5.34 to 8.39] | 5.44 [4.98 to 6.44] | 6.1 [5.6 to 7.5] | 5.9 [4.72 to 6.9] | 10.1 [9.9 to 11.8]
  WBC (1000/cubic mm)- 112: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 20 | 3
  WBC (1000/cubic mm)- 112 | 6.23 [5.1 to 6.7] | 6.39 [5.71 to 7.7] | 6.67 [5.44 to 7.98] | 5.4 [4.34 to 6.21] | 5.85 [5.09 to 6.7] | 6 [5.05 to 7.78] | 9.7 [8.9 to 10.1]
  WBC (1000/cubic mm)- 168: number analyzed (Participants) | 16 | 18 | 18 | 20 | 18 | 19 | 3
  WBC (1000/cubic mm)- 168 | 5.81 [4.61 to 7.1] | 5.51 [5.2 to 5.96] | 6.03 [5.25 to 7.6] | 5.28 [4.6 to 7.33] | 5.87 [4.71 to 7.01] | 5.7 [4.7 to 7.47] | 8.9 [8.7 to 10.9]
  WBC (1000/cubic mm)- 224: number analyzed (Participants) | 16 | 17 | 20 | 19 | 19 | 20 | 3
  WBC (1000/cubic mm)- 224 | 6.5 [4.47 to 6.8] | 5.93 [5.17 to 6.7] | 6.35 [4.88 to 7.52] | 5.3 [4.32 to 6] | 6 [5.2 to 6.6] | 5.4 [4.42 to 7.62] | 8.8 [7.2 to 11.3]
  WBC (1000/cubic mm)- 280: number analyzed (Participants) | 14 | 17 | 17 | 19 | 18 | 19 | 2
  WBC (1000/cubic mm)- 280 | 6.26 [5.3 to 7.18] | 6.59 [5.6 to 7.21] | 7 [5.13 to 7.5] | 5.56 [4.9 to 6.3] | 6.4 [5 to 7.3] | 5.8 [4.55 to 6.83] | 8.7 [7.2 to 10.2]
  WBC (1000/cubic mm)- 336: number analyzed (Participants) | 15 | 17 | 18 | 19 | 16 | 17 | 3
  WBC (1000/cubic mm)- 336 | 5.39 [4.3 to 7.57] | 6 [4.95 to 6.84] | 7.04 [5.74 to 8.4] | 5.43 [4.3 to 6.1] | 5.76 [5.37 to 6.39] | 5.49 [4.7 to 6.13] | 8.8 [8.6 to 12.1]
  WBC (1000/cubic mm)- 392: number analyzed (Participants) | 14 | 15 | 17 | 18 | 17 | 17 | 3
  WBC (1000/cubic mm)- 392 | 5.43 [4.4 to 6.9] | 5.9 [5.53 to 7.03] | 6.6 [5.29 to 7.31] | 5.08 [4.4 to 5.93] | 6.13 [5.2 to 7.5] | 5.6 [4.9 to 6.35] | 9.5 [8.5 to 9.9]
  WBC (1000/cubic mm)- 448: number analyzed (Participants) | 13 | 16 | 16 | 17 | 15 | 17 | 3
  WBC (1000/cubic mm)- 448 | 5.66 [4.6 to 6.6] | 6.26 [5.35 to 7.3] | 6 [5.23 to 8.22] | 5.45 [4.66 to 6.71] | 6.7 [4.45 to 7.1] | 5.7 [4.46 to 7] | 8.6 [8.5 to 10.6]
  WBC (1000/cubic mm)- 504: number analyzed (Participants) | 12 | 16 | 12 | 16 | 12 | 17 | 3
  WBC (1000/cubic mm)- 504 | 5.67 [4.51 to 6.65] | 6.3 [5.32 to 7.28] | 6.32 [5.2 to 8.91] | 5.55 [4.4 to 6.16] | 6.16 [5.51 to 6.7] | 5.05 [4 to 6.2] | 8.7 [8.2 to 11.9]
  WBC (1000/cubic mm)- 728: number analyzed (Participants) | 1 | 7 | 4 | 6 | 4 | 4 | 1
  WBC (1000/cubic mm)- 728 | 7.12 [7.12 to 7.12] | 6.6 [5 to 7.39] | 7.02 [5.52 to 56.95] | 4.8 [3.86 to 6] | 6.6 [6.15 to 7] | 6.18 [5.8 to 7.08] | 9.3 [9.3 to 9.3]
  Platelets (1000/cubic mm)- Screening | 260 [234.9 to 295.1] | 251 [233.6 to 265] | 271 [228 to 328.3] | 273 [209.8 to 332] | 244.5 [214.5 to 289.5] | 240.1 [223.1 to 276] | 315 [246 to 334]
  Platelets (1000/cubic mm)- 0/Enrollment: number analyzed (Participants) | 19 | 19 | 21 | 20 | 20 | 21 | 3
  Platelets (1000/cubic mm)- 0/Enrollment | 254.9 [229.1 to 291.1] | 239 [224 to 274] | 254 [219 to 317] | 270 [207.95 to 313.5] | 247 [210.5 to 281.75] | 244.5 [221 to 275] | 283 [249 to 294]
  Platelets (1000/cubic mm)- 56: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 21 | 3
  Platelets (1000/cubic mm)- 56 | 262.65 [235 to 278.7] | 255 [244 to 273] | 275.5 [238.5 to 346.1] | 283 [201 to 309] | 246 [218 to 293] | 246 [217 to 272.4] | 326 [284 to 337]
  Platelets (1000/cubic mm)- 112: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 20 | 3
  Platelets (1000/cubic mm)- 112 | 244.45 [221 to 276] | 250 [231 to 268] | 284.5 [252.5 to 337.65] | 267 [196 to 303] | 252.8 [204 to 283] | 261.5 [209.55 to 286.8] | 316 [279 to 338]
  Platelets (1000/cubic mm)- 168: number analyzed (Participants) | 16 | 18 | 18 | 20 | 18 | 19 | 3
  Platelets (1000/cubic mm)- 168 | 255.5 [234.65 to 269.05] | 255.5 [229 to 282] | 278.5 [242 to 311] | 271 [202.2 to 319.5] | 240.5 [203 to 299] | 257 [205.7 to 280] | 303 [302 to 328]
  Platelets (1000/cubic mm)- 224: number analyzed (Participants) | 16 | 17 | 20 | 19 | 19 | 20 | 3
  Platelets (1000/cubic mm)- 224 | 264 [227.5 to 277.95] | 252 [228 to 277] | 283 [250.5 to 348.5] | 252 [198 to 324] | 234 [195 to 303] | 256.5 [205.15 to 281.1] | 341 [288 to 350]
  Platelets (1000/cubic mm)- 280: number analyzed (Participants) | 14 | 17 | 17 | 19 | 18 | 19 | 2
  Platelets (1000/cubic mm)- 280 | 252.9 [229.6 to 303] | 249 [221 to 278] | 278 [222 to 338] | 250 [195 to 333] | 254.45 [215 to 287] | 257 [209 to 303.3] | 284.5 [243 to 326]
  Platelets (1000/cubic mm)- 336: number analyzed (Participants) | 15 | 17 | 18 | 19 | 16 | 17 | 3
  Platelets (1000/cubic mm)- 336 | 242 [210 to 275] | 246 [217 to 277] | 270.5 [246 to 314] | 256 [193 to 348] | 238.5 [200 to 293.15] | 233 [206.3 to 259] | 310 [286 to 324]
  Platelets (1000/cubic mm)- 392: number analyzed (Participants) | 14 | 15 | 17 | 18 | 17 | 17 | 3
  Platelets (1000/cubic mm)- 392 | 255.85 [234.6 to 282] | 255.5 [237 to 283] | 265 [244 to 311] | 251 [181 to 332] | 252 [213 to 294] | 250 [210.5 to 279.1] | 319 [283 to 321]
  Platelets (1000/cubic mm)- 448: number analyzed (Participants) | 13 | 16 | 16 | 17 | 15 | 17 | 3
  Platelets (1000/cubic mm)- 448 | 249 [241 to 276.8] | 243.5 [233 to 272.5] | 264 [223.5 to 306] | 260 [212 to 300] | 254.4 [188 to 308] | 255 [214.7 to 296] | 336 [293 to 346]
  Platelets (1000/cubic mm)- 504: number analyzed (Participants) | 12 | 16 | 12 | 16 | 12 | 17 | 3
  Platelets (1000/cubic mm)- 504 | 271.35 [244.5 to 289.6] | 252.65 [234.75 to 285] | 257.5 [246 to 338] | 268.5 [210.05 to 296] | 248.5 [193.5 to 280.5] | 251 [208.2 to 284] | 323 [251 to 325]
  Platelets (1000/cubic mm)- 728: number analyzed (Participants) | 1 | 7 | 4 | 6 | 4 | 4 | 1
  Platelets (1000/cubic mm)- 728 | 283.2 [283.2 to 283.2] | 278 [210.4 to 297] | 250 [208 to 283] | 233 [191 to 249] | 263.5 [243.95 to 295.5] | 302 [273.5 to 382.5] | 327 [327 to 327]

9. Primary Outcome: Number of Lab Grade >= 1 for Alanine Aminotransferase (ALT), Creatinine, Hemoglobin, Lymphocyte Count, Neutrophil Count, Platelets, White Blood Cells (WBC).
Description: The number (percentage) of participants with lab grade >= 1 for alanine aminotransferase (ALT), creatinine, hemoglobin, lymphocyte count, neutrophil count, platelets, white blood cells (WBC) was summarized by arm
Time Frame: Measured during screening, Days 0, 56, 112, 168, 224, 280, 336, 392, 448, 504, 728
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine | Group 7: Placebo
Number analyzed (Participants) | 19 | 19 | 21 | 21 | 20 | 21 | 3
Participants
  WBC (1000/cubic mm)- Screening | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- 0/Enrollment: number analyzed (Participants) | 19 | 19 | 21 | 20 | 20 | 21 | 3
  WBC (1000/cubic mm)- 0/Enrollment | 0 | 1 | 0 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- 56: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 21 | 3
  WBC (1000/cubic mm)- 56 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- 112: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 20 | 3
  WBC (1000/cubic mm)- 112 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- 168: number analyzed (Participants) | 16 | 18 | 18 | 20 | 18 | 19 | 3
  WBC (1000/cubic mm)- 168 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- 224: number analyzed (Participants) | 16 | 17 | 20 | 19 | 19 | 20 | 3
  WBC (1000/cubic mm)- 224 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- 280: number analyzed (Participants) | 14 | 17 | 17 | 19 | 18 | 19 | 2
  WBC (1000/cubic mm)- 280 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- 336: number analyzed (Participants) | 15 | 17 | 18 | 19 | 16 | 17 | 3
  WBC (1000/cubic mm)- 336 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- 392: number analyzed (Participants) | 14 | 15 | 17 | 18 | 17 | 17 | 3
  WBC (1000/cubic mm)- 392 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- 448: number analyzed (Participants) | 13 | 16 | 16 | 17 | 15 | 17 | 3
  WBC (1000/cubic mm)- 448 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- 504: number analyzed (Participants) | 12 | 16 | 12 | 16 | 12 | 17 | 3
  WBC (1000/cubic mm)- 504 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- 728: number analyzed (Participants) | 1 | 7 | 4 | 6 | 4 | 4 | 1
  WBC (1000/cubic mm)- 728 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- Screening | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- 0/Enrollment: number analyzed (Participants) | 19 | 19 | 21 | 20 | 20 | 21 | 3
  Neutrophils (1000/cubic mm)- 0/Enrollment | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- 56: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 21 | 3
  Neutrophils (1000/cubic mm)- 56 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- 112: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 20 | 3
  Neutrophils (1000/cubic mm)- 112 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- 168: number analyzed (Participants) | 16 | 18 | 18 | 20 | 18 | 19 | 3
  Neutrophils (1000/cubic mm)- 168 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- 224: number analyzed (Participants) | 15 | 17 | 20 | 18 | 19 | 20 | 3
  Neutrophils (1000/cubic mm)- 224 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- 280: number analyzed (Participants) | 14 | 17 | 17 | 19 | 18 | 19 | 2
  Neutrophils (1000/cubic mm)- 280 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- 336: number analyzed (Participants) | 15 | 17 | 18 | 19 | 16 | 17 | 3
  Neutrophils (1000/cubic mm)- 336 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- 392: number analyzed (Participants) | 14 | 15 | 17 | 18 | 17 | 17 | 3
  Neutrophils (1000/cubic mm)- 392 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- 448: number analyzed (Participants) | 13 | 16 | 16 | 17 | 15 | 17 | 3
  Neutrophils (1000/cubic mm)- 448 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- 504: number analyzed (Participants) | 12 | 16 | 12 | 16 | 12 | 17 | 3
  Neutrophils (1000/cubic mm)- 504 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- 728: number analyzed (Participants) | 1 | 7 | 4 | 5 | 4 | 4 | 1
  Neutrophils (1000/cubic mm)- 728 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- Screening | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- 0/Enrollment: number analyzed (Participants) | 19 | 19 | 21 | 20 | 20 | 21 | 3
  Hemoglobin (g/dL)- 0/Enrollment | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- 56: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 21 | 3
  Hemoglobin (g/dL)- 56 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- 112: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 20 | 3
  Hemoglobin (g/dL)- 112 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- 168: number analyzed (Participants) | 16 | 18 | 18 | 20 | 18 | 19 | 3
  Hemoglobin (g/dL)- 168 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- 224: number analyzed (Participants) | 16 | 17 | 20 | 19 | 19 | 20 | 3
  Hemoglobin (g/dL)- 224 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- 280: number analyzed (Participants) | 14 | 17 | 17 | 19 | 18 | 19 | 2
  Hemoglobin (g/dL)- 280 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- 336: number analyzed (Participants) | 15 | 17 | 18 | 19 | 16 | 17 | 3
  Hemoglobin (g/dL)- 336 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- 392: number analyzed (Participants) | 14 | 15 | 17 | 18 | 17 | 17 | 3
  Hemoglobin (g/dL)- 392 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- 448: number analyzed (Participants) | 13 | 16 | 16 | 17 | 15 | 17 | 3
  Hemoglobin (g/dL)- 448 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- 504: number analyzed (Participants) | 12 | 16 | 12 | 16 | 12 | 17 | 3
  Hemoglobin (g/dL)- 504 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- 728: number analyzed (Participants) | 1 | 7 | 4 | 6 | 4 | 4 | 1
  Hemoglobin (g/dL)- 728 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- Screening | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- 0/Enrollment: number analyzed (Participants) | 19 | 19 | 21 | 20 | 20 | 21 | 3
  Lymphocytes (1000/cubic mm)- 0/Enrollment | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- 56: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 21 | 3
  Lymphocytes (1000/cubic mm)- 56 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- 112: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 20 | 3
  Lymphocytes (1000/cubic mm)- 112 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- 168: number analyzed (Participants) | 16 | 18 | 18 | 20 | 18 | 19 | 3
  Lymphocytes (1000/cubic mm)- 168 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- 224: number analyzed (Participants) | 15 | 17 | 20 | 18 | 19 | 20 | 3
  Lymphocytes (1000/cubic mm)- 224 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- 280: number analyzed (Participants) | 14 | 17 | 17 | 19 | 18 | 19 | 2
  Lymphocytes (1000/cubic mm)- 280 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- 336: number analyzed (Participants) | 15 | 17 | 18 | 19 | 16 | 17 | 3
  Lymphocytes (1000/cubic mm)- 336 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- 392: number analyzed (Participants) | 14 | 15 | 17 | 18 | 17 | 17 | 3
  Lymphocytes (1000/cubic mm)- 392 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- 448: number analyzed (Participants) | 13 | 16 | 16 | 17 | 15 | 17 | 3
  Lymphocytes (1000/cubic mm)- 448 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- 504: number analyzed (Participants) | 12 | 16 | 12 | 16 | 12 | 17 | 3
  Lymphocytes (1000/cubic mm)- 504 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- 728: number analyzed (Participants) | 1 | 7 | 4 | 5 | 4 | 4 | 1
  Lymphocytes (1000/cubic mm)- 728 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Screening | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- 0/Enrollment: number analyzed (Participants) | 19 | 19 | 21 | 20 | 20 | 21 | 3
  Platelets (1000/cubic mm)- 0/Enrollment | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- 56: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 21 | 3
  Platelets (1000/cubic mm)- 56 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- 112: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 20 | 3
  Platelets (1000/cubic mm)- 112 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- 168: number analyzed (Participants) | 16 | 18 | 18 | 20 | 18 | 19 | 3
  Platelets (1000/cubic mm)- 168 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- 224: number analyzed (Participants) | 16 | 17 | 20 | 19 | 19 | 20 | 3
  Platelets (1000/cubic mm)- 224 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- 280: number analyzed (Participants) | 14 | 17 | 17 | 19 | 18 | 19 | 2
  Platelets (1000/cubic mm)- 280 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- 336: number analyzed (Participants) | 15 | 17 | 18 | 19 | 16 | 17 | 3
  Platelets (1000/cubic mm)- 336 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- 392: number analyzed (Participants) | 14 | 15 | 17 | 18 | 17 | 17 | 3
  Platelets (1000/cubic mm)- 392 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- 448: number analyzed (Participants) | 13 | 16 | 16 | 17 | 15 | 17 | 3
  Platelets (1000/cubic mm)- 448 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Platelets (1000/cubic mm)- 504: number analyzed (Participants) | 12 | 16 | 12 | 16 | 12 | 17 | 3
  Platelets (1000/cubic mm)- 504 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- 728: number analyzed (Participants) | 1 | 7 | 4 | 6 | 4 | 4 | 1
  Platelets (1000/cubic mm)- 728 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Screening | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)- 0/Enrollment: number analyzed (Participants) | 19 | 19 | 21 | 20 | 20 | 21 | 3
  ALT (SGPT) (U/L)- 0/Enrollment | 0 | 0 | 0 | 0 | 1 | 1 | 0
  ALT (SGPT) (U/L)- 56: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 21 | 3
  ALT (SGPT) (U/L)- 56 | 0 | 0 | 2 | 0 | 0 | 0 | 1
  ALT (SGPT) (U/L)- 112: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 20 | 3
  ALT (SGPT) (U/L)- 112 | 0 | 0 | 1 | 0 | 2 | 1 | 1
  ALT (SGPT) (U/L)- 168: number analyzed (Participants) | 16 | 18 | 18 | 20 | 18 | 19 | 3
  ALT (SGPT) (U/L)- 168 | 1 | 1 | 1 | 1 | 1 | 1 | 1
  ALT (SGPT) (U/L)- 224: number analyzed (Participants) | 16 | 17 | 20 | 19 | 19 | 20 | 3
  ALT (SGPT) (U/L)- 224 | 1 | 0 | 0 | 0 | 1 | 0 | 1
  ALT (SGPT) (U/L)- 280: number analyzed (Participants) | 14 | 17 | 17 | 19 | 19 | 19 | 2
  ALT (SGPT) (U/L)- 280 | 1 | 0 | 0 | 2 | 1 | 1 | 0
  ALT (SGPT) (U/L)- 336: number analyzed (Participants) | 15 | 17 | 18 | 19 | 16 | 17 | 3
  ALT (SGPT) (U/L)- 336 | 0 | 0 | 0 | 1 | 0 | 1 | 1
  ALT (SGPT) (U/L)- 392: number analyzed (Participants) | 14 | 15 | 17 | 18 | 17 | 17 | 3
  ALT (SGPT) (U/L)- 392 | 3 | 0 | 0 | 0 | 0 | 0 | 1
  ALT (SGPT) (U/L)- 448: number analyzed (Participants) | 13 | 16 | 16 | 17 | 15 | 17 | 3
  ALT (SGPT) (U/L)- 448 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  ALT (SGPT) (U/L)- 504: number analyzed (Participants) | 12 | 16 | 12 | 16 | 12 | 17 | 3
  ALT (SGPT) (U/L)- 504 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  ALT (SGPT) (U/L)- 728: number analyzed (Participants) | 1 | 7 | 4 | 6 | 4 | 4 | 1
  ALT (SGPT) (U/L)- 728 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL)- Screening | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL)- 0/Enrollment: number analyzed (Participants) | 19 | 19 | 21 | 20 | 19 | 21 | 3
  Creatinine (mg/dL)- 0/Enrollment | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Creatinine (mg/dL)- 56: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 21 | 3
  Creatinine (mg/dL)- 56 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL)- 112: number analyzed (Participants) | 18 | 18 | 20 | 21 | 19 | 20 | 3
  Creatinine (mg/dL)- 112 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Creatinine (mg/dL)- 168: number analyzed (Participants) | 16 | 18 | 18 | 20 | 18 | 19 | 3
  Creatinine (mg/dL)- 168 | 0 | 0 | 0 | 2 | 0 | 1 | 0
  Creatinine (mg/dL)- 224: number analyzed (Participants) | 16 | 17 | 20 | 19 | 19 | 20 | 3
  Creatinine (mg/dL)- 224 | 0 | 0 | 1 | 1 | 1 | 0 | 0
  Creatinine (mg/dL)- 280: number analyzed (Participants) | 14 | 17 | 17 | 19 | 19 | 19 | 2
  Creatinine (mg/dL)- 280 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Creatinine (mg/dL)- 336: number analyzed (Participants) | 15 | 17 | 18 | 19 | 16 | 17 | 3
  Creatinine (mg/dL)- 336 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Creatinine (mg/dL)- 392: number analyzed (Participants) | 14 | 15 | 17 | 18 | 17 | 17 | 3
  Creatinine (mg/dL)- 392 | 0 | 0 | 0 | 2 | 3 | 0 | 0
  Creatinine (mg/dL)- 448: number analyzed (Participants) | 13 | 16 | 16 | 17 | 15 | 17 | 3
  Creatinine (mg/dL)- 448 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Creatinine (mg/dL)- 504: number analyzed (Participants) | 12 | 16 | 12 | 16 | 12 | 17 | 3
  Creatinine (mg/dL)- 504 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Creatinine (mg/dL)- 728: number analyzed (Participants) | 1 | 7 | 4 | 6 | 4 | 4 | 1
  Creatinine (mg/dL)- 728 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: VRC07523LS Serum Concentrations
Description: VRC07523LS serum concentrations measured in healthy human subjects after up to five administrations of the study product via the IV, SC or IM routes at various doses. Serum concentrations between the first and second study product administrations (Target Visit Day 0-112) were measured using ELISA assay in all enrolled participants. Serum concentrations after the second study product administrations (Target Visit Day 168-784) were measured using BAMA (LUMINEX) assay in a subset of participants enrolled in each treatment group and all particiants in plocebo group. serum concentrations below the lower limit of quantification (LLoQ) were replaced by half the LLoQ. Thus, concentrations below the LLoQ when measured by the ELISA assay were replaced by 0.5 ug/ml and concentrations below the LLoQ when measured by the BAMA assay were replaced by 0.02285 ug/ml.
Time Frame: Target Visit Days 0, 3, 6, 28, 56, 84, 112, 168, 224, 280, 336, 392, 448, 504, 560, 616, 672, 728, 784 (i.e., visit numbers 2 through 20)
Population: Overall Number of Participants Analyzed represents the number of enrolled participants. Number Analyzed shows the number of participants with available data after filtering for assay specific quality control criteria at each timepoint.
Measure: Median (Inter-Quartile Range); unit: ug/ml
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine | Group 7: Placebo
Number analyzed (Participants) | 19 | 19 | 21 | 21 | 20 | 21 | 3
ug/ml
  IDVRC07-523LS (Day-000): number analyzed (Participants) | 18 | 17 | 19 | 20 | 19 | 20 | 3
  IDVRC07-523LS (Day-000) | 0.5 [0.5 to 0.5] | 0.5 [0.5 to 0.5] | 0.5 [0.5 to 0.5] | 0.5 [0.5 to 0.5] | 0.5 [0.5 to 0.5] | 0.5 [0.5 to 0.5] | 0.5 [0.5 to 0.5]
  IDVRC07-523LS (Day-003): number analyzed (Participants) | 17 | 16 | 20 | 20 | 18 | 20 | 2
  IDVRC07-523LS (Day-003) | 43.13 [38.57 to 52.81] | 80.7 [73.52 to 101.15] | 332.57 [260 to 455.77] | 11.06 [7.95 to 15.28] | 17.81 [14.57 to 26.49] | 16.71 [15.16 to 19.14] | 0.5 [0.5 to 0.5]
  IDVRC07-523LS (Day-006): number analyzed (Participants) | 18 | 17 | 19 | 18 | 18 | 20 | 3
  IDVRC07-523LS (Day-006) | 27.71 [23.7 to 33.64] | 59.05 [49.91 to 71.34] | 224 [200.96 to 261.88] | 11.04 [8.26 to 13.21] | 22.22 [18.81 to 26.26] | 16.03 [13.89 to 17.81] | 0.5 [0.5 to 0.5]
  IDVRC07-523LS (Day-028): number analyzed (Participants) | 18 | 17 | 20 | 20 | 18 | 20 | 3
  IDVRC07-523LS (Day-028) | 14.56 [13.48 to 17.86] | 27.86 [25.92 to 36.53] | 125.17 [110.6 to 132.2] | 6.79 [5.63 to 8.36] | 13.37 [11.89 to 17.65] | 10.03 [8.91 to 11.87] | 0.5 [0.5 to 0.5]
  IDVRC07-523LS (Day-056): number analyzed (Participants) | 18 | 17 | 19 | 20 | 18 | 20 | 3
  IDVRC07-523LS (Day-056) | 10.67 [8.26 to 12.76] | 17.08 [15.32 to 21.55] | 68.97 [59.45 to 75.21] | 5.02 [3.81 to 5.7] | 7.63 [6.57 to 10.43] | 6.27 [5.72 to 7.39] | 0.5 [0.5 to 0.5]
  IDVRC07-523LS (Day-084): number analyzed (Participants) | 18 | 16 | 19 | 18 | 16 | 19 | 3
  IDVRC07-523LS (Day-084) | 5.43 [4.69 to 6.9] | 12.19 [10.33 to 14.17] | 45.27 [36.41 to 52.23] | 2.99 [0.86 to 4.12] | 5.9 [4.89 to 7.23] | 4.29 [3.48 to 5.33] | 0.5 [0.5 to 0.5]
  IDVRC07-523LS (Day-112): number analyzed (Participants) | 18 | 17 | 20 | 20 | 19 | 20 | 3
  IDVRC07-523LS (Day-112) | 4.08 [3.09 to 4.84] | 6.51 [5.33 to 7.59] | 26.83 [22.83 to 30.69] | 0.5 [0.5 to 2.14] | 3.95 [2.72 to 4.58] | 2.98 [1.88 to 3.53] | 0.5 [0.5 to 0.5]
  IDVRC07-523LS (Day-168): number analyzed (Participants) | 9 | 9 | 9 | 8 | 9 | 11 | 3
  IDVRC07-523LS (Day-168) | 13.14 [8.75 to 14.82] | 22.46 [19.66 to 24.95] | 98.34 [93.59 to 111.17] | 5.77 [4.19 to 6.56] | 10.99 [10.15 to 12.2] | 8.09 [6.07 to 8.74] | 0.02 [0.02 to 0.02]
  IDVRC07-523LS (Day-224): number analyzed (Participants) | 9 | 9 | 10 | 9 | 10 | 11 | 3
  IDVRC07-523LS (Day-224) | 5.55 [5.12 to 7.08] | 9.83 [8.89 to 11.74] | 36.11 [29.29 to 49.15] | 2.31 [1.11 to 3.17] | 5.95 [4.95 to 7.17] | 3.53 [2.41 to 4.52] | 0.02 [0.02 to 0.02]
  IDVRC07-523LS (Day-280): number analyzed (Participants) | 9 | 9 | 10 | 9 | 10 | 11 | 2
  IDVRC07-523LS (Day-280) | 12.17 [11.3 to 14.1] | 25.77 [20.13 to 27.8] | 93.35 [81.62 to 100.24] | 7.52 [3.42 to 8.66] | 13.65 [10.92 to 17.55] | 7.79 [5.88 to 10.33] | 0.02 [0.02 to 0.02]
  IDVRC07-523LS (Day-336): number analyzed (Participants) | 9 | 9 | 10 | 9 | 10 | 11 | 3
  IDVRC07-523LS (Day-336) | 5.5 [3.8 to 6.52] | 11.15 [7.74 to 12.77] | 38.01 [25.6 to 48.67] | 2.16 [1.49 to 3.2] | 6.39 [4.86 to 8.61] | 3.62 [2.82 to 4.01] | 0.02 [0.02 to 0.02]
  IDVRC07-523LS (Day-392): number analyzed (Participants) | 9 | 8 | 10 | 9 | 10 | 11 | 3
  IDVRC07-523LS (Day-392) | 13.31 [10.04 to 14.6] | 25.88 [22.09 to 30.52] | 98.93 [86.92 to 113.48] | 6.12 [3.94 to 8.47] | 12.76 [11.08 to 15.29] | 8.13 [6.66 to 9.47] | 0.02 [0.02 to 0.02]
  IDVRC07-523LS (Day-448): number analyzed (Participants) | 9 | 9 | 10 | 9 | 10 | 11 | 3
  IDVRC07-523LS (Day-448) | 5.6 [4.24 to 6.81] | 10.29 [9.04 to 15.12] | 40.22 [36.47 to 46.45] | 2.71 [2 to 4.39] | 6.06 [5.28 to 6.88] | 3.59 [3.23 to 4.26] | 0.02 [0.02 to 0.02]
  IDVRC07-523LS (Day-504): number analyzed (Participants) | 9 | 9 | 10 | 9 | 10 | 11 | 3
  IDVRC07-523LS (Day-504) | 14.18 [8.37 to 14.92] | 23.4 [20.28 to 28.7] | 98.2 [93.78 to 106.21] | 6.11 [4.77 to 8.11] | 13.22 [10.63 to 15.47] | 7.61 [6.58 to 8.92] | 0.02 [0.02 to 0.02]
  IDVRC07-523LS (Day-560): number analyzed (Participants) | 8 | 7 | 6 | 7 | 8 | 7 | 3
  IDVRC07-523LS (Day-560) | 5.08 [3.62 to 6.69] | 10.67 [9.21 to 15.27] | 41.17 [32.3 to 49.84] | 1.65 [1.42 to 3.68] | 7.17 [6.18 to 8.09] | 3.92 [3.56 to 4.32] | 0.02 [0.02 to 0.02]
  IDVRC07-523LS (Day-616): number analyzed (Participants) | 6 | 5 | 6 | 9 | 4 | 4 | 0
  IDVRC07-523LS (Day-616) | 2.7 [2.36 to 3.68] | 5.74 [4.59 to 6.72] | 20.78 [16.32 to 27.46] | 1.52 [0.58 to 1.96] | 3.63 [2.8 to 3.83] | 1.36 [0.89 to 1.69] |
  IDVRC07-523LS (Day-672): number analyzed (Participants) | 5 | 8 | 4 | 5 | 8 | 2 | 0
  IDVRC07-523LS (Day-672) | 1.14 [0.95 to 1.18] | 2.81 [1.67 to 3.63] | 10.68 [9.02 to 11.7] | 0.78 [0.61 to 1.45] | 1.29 [0.91 to 1.52] | 1.25 [0.95 to 1.56] |
  IDVRC07-523LS (Day-728): number analyzed (Participants) | 4 | 5 | 5 | 5 | 6 | 4 | 2
  IDVRC07-523LS (Day-728) | 0.47 [0.33 to 0.62] | 1.68 [0.59 to 2.27] | 5.87 [3.11 to 5.94] | 0.45 [0.45 to 0.85] | 0.74 [0.69 to 0.83] | 0.44 [0.33 to 0.47] | 0.02 [0.02 to 0.02]
  IDVRC07-523LS (Day-784): number analyzed (Participants) | 7 | 4 | 9 | 8 | 7 | 9 | 3
  IDVRC07-523LS (Day-784) | 0.51 [0.26 to 0.54] | 0.94 [0.72 to 1.09] | 2.17 [1.76 to 3.01] | 0.17 [0.1 to 0.33] | 0.36 [0.34 to 0.52] | 0.27 [0.2 to 0.29] | 0.02 [0.02 to 0.02]

11. Secondary Outcome: Occurrence of Antidrug Antibodies (ADA)
Description: Antidrug antibodies (ADA) are most typically detected and characterized using a tiered testing strategy. In Tier I, a sensitive binding assay is used to determine if samples may have ADA present. In Tier II, the response is confirmed, typically by establishing the specificity of the response by competition with free drug. In Tier III, the response is characterized, typically with a neutralization reduction assay and/or a titering assay.
Time Frame: Day 0, 6, 112, 224, 448
Population: Overall Number of Participants Analyzed presents the number of enrolled participants in each treatment arm. Number Analyzed shows the number of samples available and tested in the certain tier and timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine | Group 7: Placebo
Number analyzed (Participants) | 19 | 19 | 21 | 21 | 20 | 21 | 3
Participants
  0 - Tier I | 2 | 2 | 0 | 2 | 0 | 1 | 0
  0 - Tier II: number analyzed (Participants) | 2 | 2 | 0 | 2 | 0 | 1 | 0
  0 - Tier II | 0 | 0 |  | 0 |  | 0 |
  0 - Tier III: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  112 - Tier I: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0 | 0
  112 - Tier I |  |  | 0 |  | 0 |  |
  112 - Tier II: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  112 - Tier III: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  224 - Tier I: number analyzed (Participants) | 16 | 17 | 20 | 19 | 19 | 20 | 3
  224 - Tier I | 0 | 0 | 0 | 1 | 0 | 0 | 0
  224 - Tier II: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  224 - Tier II |  |  |  | 1 |  |  |
  224 - Tier III: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  224 - Tier III |  |  |  | 0 |  |  |
  448 - Tier I: number analyzed (Participants) | 13 | 15 | 16 | 17 | 15 | 17 | 3
  448 - Tier I | 0 | 1 | 0 | 0 | 0 | 0 | 0
  448 - Tier II: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  448 - Tier II |  | 0 |  |  |  |  |
  448 - Tier III: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  6 - Tier I: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  6 - Tier I |  | 0 |  |  |  |  |
  6 - Tier II: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  6 - Tier III: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Magnitude and Breadth of Neutralizing Antibody Responses Against Autologous Viral Isolates as Assessed by Area Under the Magnitude-breadth Curves 8, 72, 88 Weeks After the First Study Product Administration.
Description: Magnitude-breadth characterize the magnitude (ID50 or ID80 titers) and breadth (number of virus isolates) of each individual serum sample assayed against a panel of virus isolates. MB curves show, for each possible magnitude threshold, the fraction of assays with magnitudes greater than this threshold. The area under the magnitude-breadth curve (AUC-MB) is calculated as the average of the log10-based ID50 or ID80 titers over the panel of isolates. Isolates includes: H703_0646_051sN, H703_1471_190s, H703_1750_140Es, H704_0726_080sN, H704_1535_030sN, H704_2544_140eN01, PVO.4.
Time Frame: Weeks 8, 72, and 88 following the first study product administration
Population: Overall Number of Participants Analyzed- represents the number of sampled participants. Number Analyzed shows the number of participants with available nAb data after filtering for assay specific quality control criteria at each timepoint.
Measure: Median (Inter-Quartile Range); unit: log10(titer)
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine
Number analyzed (Participants) | 19 | 19 | 21 | 21 | 20 | 21
log10(titer)
  ID50 (Week-08): number analyzed (Participants) | 9 | 10 | 10 | 10 | 10 | 11
  ID50 (Week-08) | 1.56 [1.44 to 1.56] | 1.89 [1.74 to 2] | 2.46 [2.38 to 2.54] | 1.34 [1.23 to 1.54] | 1.54 [1.4 to 1.55] | 1.39 [1.26 to 1.45]
  ID50 (Week-72): number analyzed (Participants) | 9 | 10 | 10 | 10 | 10 | 11
  ID50 (Week-72) | 1.62 [1.57 to 1.81] | 2.03 [1.79 to 2.12] | 2.6 [2.5 to 2.67] | 1.36 [1.25 to 1.55] | 1.6 [1.48 to 1.71] | 1.49 [1.42 to 1.57]
  ID50 (Week-88): number analyzed (Participants) | 6 | 5 | 6 | 10 | 4 | 3
  ID50 (Week-88) | 0.98 [0.96 to 1.11] | 1.4 [1.26 to 1.4] | 1.93 [1.85 to 2.07] | 0.8 [0.7 to 0.94] | 0.97 [0.89 to 0.98] | 0.9 [0.8 to 0.96]
  ID80 (Week-08): number analyzed (Participants) | 9 | 10 | 10 | 10 | 10 | 11
  ID80 (Week-08) | 1.14 [1.04 to 1.19] | 1.37 [1.33 to 1.42] | 1.97 [1.89 to 2.03] | 0.93 [0.89 to 1.11] | 1.15 [1.03 to 1.2] | 1.01 [0.91 to 1.08]
  ID80 (Week-72): number analyzed (Participants) | 9 | 10 | 10 | 10 | 10 | 11
  ID80 (Week-72) | 1.27 [1.16 to 1.33] | 1.49 [1.35 to 1.55] | 2.14 [2.02 to 2.16] | 1 [0.88 to 1.12] | 1.21 [1.12 to 1.29] | 1.13 [1.02 to 1.18]
  ID80 (Week-88): number analyzed (Participants) | 6 | 5 | 6 | 10 | 4 | 3
  ID80 (Week-88) | 0.85 [0.77 to 0.88] | 0.91 [0.88 to 0.95] | 1.45 [1.41 to 1.55] | 0.7 [0.7 to 0.74] | 0.84 [0.8 to 0.84] | 0.75 [0.72 to 0.79]

ADVERSE EVENTS:
Time Frame: The study Unsolicited AE reporting time frame is from study enrollment of a trial participant to (and including) the Week 112 visit (v20.0). The Solicited AE assessment were collected through 3 full days after each vaccination (vaccinations were given at weeks 0, 16, 32, 48 and 64).
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine | Group 7: Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/21 | 0/21 | 0/20 | 0/21 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/19 | 1/19 | 0/21 | 1/21 | 0/20 | 0/21 | 0/3
Other Adverse Events (participants affected / at risk) | 14/19 | 16/19 | 14/21 | 18/21 | 16/20 | 17/21 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Vaccine (N=19) | Group 2: Vaccine (N=19) | Group 3: Vaccine (N=21) | Group 4: Vaccine (N=21) | Group 5: Vaccine (N=20) | Group 6: Vaccine (N=21) | Group 7: Placebo (N=3)
Any Event in SOC (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Vaccine (N=19) | Group 2: Vaccine (N=19) | Group 3: Vaccine (N=21) | Group 4: Vaccine (N=21) | Group 5: Vaccine (N=20) | Group 6: Vaccine (N=21) | Group 7: Placebo (N=3)
Any Event in SOC (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mitral valve prolapse (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eczema eyelids (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid rash (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Gastrointestinal disorders) | 1 (1) | 7 (8) | 5 (5) | 2 (3) | 6 (7) | 3 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Plicated tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (General disorders) | 3 (3) | 3 (4) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Infections and infestations) | 9 (12) | 10 (31) | 11 (27) | 9 (15) | 10 (14) | 12 (21) | 3 (9)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Anorectal human papilloma virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial vulvovaginitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 5 (9) | 7 (10) | 3 (4) | 4 (5) | 6 (7) | 3 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (5) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 2 (2) | 3 (7) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Viral pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Any Event in SOC (Injury, poisoning and procedural complications) | 3 (4) | 4 (4) | 4 (7) | 4 (6) | 4 (4) | 4 (4) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Investigations) | 4 (7) | 3 (5) | 8 (15) | 9 (19) | 5 (11) | 5 (7) | 2 (6)
Alanine aminotransferase abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (5) | 1 (2) | 3 (4) | 3 (4) | 2 (4) | 2 (3) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 3 (3) | 5 (8) | 3 (4) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 1 (2) | 2 (3) | 1 (4) | 1 (1) | 2 (2) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Red blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Smear cervix abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Any Event in SOC (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (6) | 1 (1) | 6 (9) | 4 (6) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteochondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 3 (4) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruxism (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burnout syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 0 (0) | 3 (3) | 3 (5) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Skin and subcutaneous tissue disorders) | 2 (3) | 4 (4) | 0 (0) | 4 (4) | 3 (3) | 1 (2) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/50/NCT03387150/Prot_SAP_000.pdf